CLINICAL TRIAL: NCT01973673
Title: Healthy Bones Study: An Intervention to Improve Healthy Bone Behaviours in Prostate Cancer Patients on Androgen Deprivation Therapy (ADT)
Brief Title: Healthy Bones Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-6050
Record Dates: First submitted 2013-09-30; First posted 2013-10-31 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Locally Advanced Malignant Neoplasm
Keywords: prostate cancer; ADT; bone health
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bone health educational materials (Active Comparator): Bone health written educational materials, Bone health prescription,verbal counselling
  Interventions: Behavioral: Bone health educational materials
- Usual care (No Intervention): Usual clinical care to be provided by oncologists.

INTERVENTIONS:
Behavioral: Bone health educational materials
  Arms: Bone health educational materials

SUMMARY:
Prostate cancer patients receiving hormone treatment (androgen deprivation therapy, or ADT) are at increased risk of developing bone loss and osteoporosis as side effects. To prevent this, guidelines recommend participation in healthy bone behaviours including weight-bearing exercise and adequate calcium/vitamin D intake. However, prior studies have shown that patients are not regularly screened or counselled regarding healthy bone behaviours while receiving ADT. Maintaining bone health in prostate cancer patients is important because men on ADT are at increased risk of fractures. In this study, the investigators will examine whether an intervention designed to improve healthy bone behaviours among prostate cancer patients on ADT can be implemented. The intervention consists of a written "healthy bones prescription", brief verbal counseling, and printed educational materials for participants. Investigators hope to obtain an initial estimate of whether the intervention works. They also hope to show that this simple intervention can be implemented in a real, working cancer clinic.

The investigators hypothesize that an intervention to improve bone health in prostate cancer patients receiving ADT (healthy bones prescription, verbal counseling, and printed educational materials) is effective, implementable, and accepted by clinicians and patients.

DETAILED DESCRIPTION:
The study has a before-and-after design, to allow comparison of the intervention before its implementation and after its implementation. This design permits a reliable assessment of baseline characteristics prior to implementation of intervention and over time, particularly in situations where randomization is not feasible (e.g. due to contamination of treating physicians). The point at which the intervention will start to be delivered for new study participants is when 150 patients are accrued to the Before arm.

1. Before/control arm (Before arm) Usual care by Princess Margaret Cancer Centre (PM) oncologist.
2. After/intervention arm (After arm) Provision of a healthy bones prescription, verbal counselling, and written educational materials regarding healthy bone behaviours by PM oncologist or delegate (e.g. clinical fellow), in addition to usual care by oncologist. The intervention may be delivered again at a subsequent follow-up at the request of the patient and/or at the discretion of the oncologist.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer patients receiving ADT at study entry (for a maximum of 12 months prior to study entry or planning to receive ADT within 3 weeks of study entry), for an expected duration of >6 months; Eastern Cooperative Oncology Group (ECOG) performance status <3

Exclusion Criteria: Unable to exercise (e.g. major physical disability, severe osteoarthritis, or other severe comorbidity); severe cardiac disease (congestive heart failure with New York Heart Association (NYHA) class >2, angioplasty/coronary artery bypass surgery within 3 months of study entry); patients with bone endocrinopathy (parathyroid disorders, osteomalacia); stage IV-V chronic kidney disease (estimated glomerular filtration rate [eGFR] <30 mL/min/1.75 m2; prior serum creatinine not required for entry into study); allergy to components of calcium & vitamin D tablets.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Proportion of eligible and consented patients who complete study follow-up, as a measure of study feasibility
Study completion and retention rate | 3 months
  Change in patient-reported daily calcium intake, as a measure of intervention efficacy
Intervention efficacy | 3 months
  Change in patient-reported weekly exercise duration, as a measure of intervention efficacy

SECONDARY OUTCOMES:
Clinical outcome | 6 months
  Proportion of patients whose calcium, vitamin D intake, and exercise may be assessed from properly completed questionnaires
Clinical outcome capture rate | 6 months
  Patient and clinician satisfaction with clinical study on a ten-point scale
Questionnaire, and Osteoporosis Health Belief Scale | 3 months
  Change in patient knowledge and health benefits regarding osteoporosis, as determined with Facts on Osteoporosis Quiz - Revised, Men's Osteoporosis Knowledge
BMD monitoring | 6 months
  Proportion of enrolled patients having bone mineral density (BMD) tests performed within 6 months of ADT initiation

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — UHN
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsang DS, Jones JM, Samadi O, Shah S, Mitsakakis N, Catton CN, Jeon W, To J, Breunis H, Alibhai SMH. Healthy Bones Study: can a prescription coupled with education improve bone health for patients receiving androgen deprivation therapy?-a before/after study. Support Care Cancer. 2018 Aug;26(8):2861-2869. doi: 10.1007/s00520-018-4150-0. Epub 2018 Mar 12. PMID 29532243